CLINICAL TRIAL: NCT01229293
Title: The Effect of Implant Design on Postoperative Mechanical Muscle Function Recovery and Gait in Hip Replacement Patients: A Randomized Clinical Trail
Brief Title: Gait Analysis and Neuromuscular Function After Primary Total Hip Replacement
Acronym: RTHA and THA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government); The Danish Rheumatism Association (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Carsten Jensen, PhD-fellow, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VF20050133-2
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis
Keywords: Mechanical muscle function; Muscle strength; Hip replacement; Osteoarthritis; Hip arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resurfacing Total Hip Arthroplasty (Experimental): A hip replacement that leaves most of the underlying bone intact and mimics the natural biomechanical features of the hip joint. Articular surface replacement ASR, DePuy posterolateral approach used (RTHA)
  Interventions: Procedure: Articular Surface Replacement (ASR)
- Standard Total Hip Arthroplasty (THA) (Active Comparator): A standard 28 mm head uncemented THA
  Interventions: Procedure: Standard Total Hip Arthroplasty (THA)

INTERVENTIONS:
Procedure: Articular Surface Replacement (ASR) — Articular surface replacement, DePuy, posterolateral approach used
  Arms: Resurfacing Total Hip Arthroplasty
Procedure: Standard Total Hip Arthroplasty (THA) — Device: Biomet 28mm
  Arms: Standard Total Hip Arthroplasty (THA)

SUMMARY:
This study is conducted at Odense University Hospital(OUH) in collaboration with Institute of Clinical Biomechanics and Sport Science, University of Southern Denmark and Clinical Institute, University of Southern Denmark

Aim: To evaluate the effect of implant design on postoperative total leg muscle function recovery and gait in hip replacement patients.

Design: A prospective randomized controlled clinical trial where patients are randomized into (A) total hip arthroplasty surgery (THA) or (B) resurfacing total hip replacement surgery (RTHA). Pre-surgery assessment and follow-up will be conducted at 8, 26 and 52 wks post-surgery.

DETAILED DESCRIPTION:
The project consist of three substudies:

* Determination of test-retest reliability and agreement of specific mechanical muscle function variables for the patients of interest.
* Evaluate the effect of implant design on postoperative mechanical muscle recovery
* Evaluate the effect of implant design on postoperative gait

ELIGIBILITY:
Inclusion Criteria:

* Primary arthrosis

Exclusion Criteria:

* Osteoporosis, (T-score < 2.5 SD) of proximal femur
* BMI > 35
* Severe acetabulum dysplasia (AP centre edge < 15-20°)
* Femur anteversion > 25°
* Severe caput deformity
* Leg length discrepancy > 1 cm
* Off-set problems
* Earlier fracture of the ipsilateral proximal femur
* Rheumatoid arthritis
* Neuromuscular or vascular disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-02; Primary Completion 2010-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Maximal muscle strength (Peak torque, Nm) | 52 wks post-surgery (primary endpoint)
  Maximal muscle strength (peak torque, Nm) during maximal voluntary unilateral knee extension-flexion (seated), hip extension-flexion, and hip adduction-abduction (standing), respectively. Both the affected (AF) and non-affected (NA) leg

SECONDARY OUTCOMES:
Rapid force capacity (Rate of torque development, Nm/sec) | 52 wks post-surgery (primary endpoint)
  Determined as the mean tangential slope of the torque-time curve in time intervals 0-100ms (RTD100ms), 0-200ms (RTD200ms) and 0-peak (RTD peak) relative to onset of contraction (t = 0ms)
Gait parameters | 26 wks post-surgery (primary endpoint)
  Selfselected, matched and maximal speed, limb index, Gait deviation index, Movement profile analysis togeter with tempo- spatial parameters
Postural Control | 52 wks post-surgery (primary endpoint)
  Sway analysis (postural control) during two-leg standing, tandem, one-leg standing and during transistion from sit-to-stand.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Overgaard, Prof., MD., PhD, Study Chair — Odense University Hospital
Locations (1):
- Orthopaedic Research Unit, Dept. of Orthopaedic Surgery and Traumatology, Odense University Hospital, Inst. of Clinical Research - University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Jensen C, Rosenlund S, Nielsen DB, Overgaard S, Holsgaard-Larsen A. The use of the Gait Deviation Index for the evaluation of participants following total hip arthroplasty: An explorative randomized trial. Gait Posture. 2015 Jun;42(1):36-41. doi: 10.1016/j.gaitpost.2015.02.009. Epub 2015 Apr 28. PMID 25957650
- [Derived] Jensen C, Aagaard P, Overgaard S. Recovery in mechanical muscle strength following resurfacing vs standard total hip arthroplasty - a randomised clinical trial. Osteoarthritis Cartilage. 2011 Sep;19(9):1108-16. doi: 10.1016/j.joca.2011.06.011. Epub 2011 Jun 28. PMID 21749928